CLINICAL TRIAL: NCT04119479
Title: Interdisziplinäre Plattform für Rehabilitationsforschung Und Innovative Versorgung Von SchlaganfallpatientInnen - ImPRoVe Interdisciplinary Platform for Rehabilitation Research and Innovative Care of Stroke Patients - ImPRoVe
Brief Title: Interdisciplinary Platform for Rehabilitation Research and Innovative Care of Stroke Patients
Acronym: ImPRoVe
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsche Rentenversicherung (Other)
Responsible Party: Sponsor
Other Study IDs: IMPROVE
Record Dates: First submitted 2019-09-26; First posted 2019-10-08 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Stroke
Keywords: Functional recovery; Neurorehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study of functional recovery of stroke patients after discharge from rehabilitation

DETAILED DESCRIPTION:
Cerebrovascular diseases, such as stroke, are among the greatest challenges in healthcare. This proves the importance of neuro-rehabilitative research. Stroke research is often focused on the acute treatment phase as well as the inpatient rehabilitation. A remaining question is how do stroke patients clinically develop after being discharged from the hospital? How stable are the achieved rehabilitation effects and how much more clinical improvement is seen in the following time period, especially with regard to ICF functionality? In this observational longitudinal study, the current practice of neurorehabilitation will be investigated and the influence of motor skills, cognition, care situation, depression, information and fatigue on functional recovery as well as participation, autonomy and quality of life will be evaluated. Stroke patients will be examined at the end of rehabilitation, after three, six and 12 months. In addition, a group of chronic patients undergoes the same examinations and thereby represents a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or haemorrhagic stroke according to ICD 10 I61-I69
* Patients in or after completion of rehabilitation phases C and D according to BAR criteria
* Age >= 18
* Sufficient knowledge of German
* Existing declaration of consent
* Deficit still existing (Rankin score of at least 1 at inclusion)

Exclusion Criteria:

* need for care prior stroke
* SAB, craniocerebral trauma, TIA as primary diagnosis
* Severe pre-existing psychiatric disease
* Participation in follow-up examination not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnoses cerebral infarction and/or cerebral hemorrhage corresponding to the diagnoses of ICD 10 I61-I69 from rehabilitation phases C and D according to the criteria of the Bundesarbeitsgemeinschaft für Rehabilitation (BAR) shall be included at the end of inpatient rehabilitation therapy. The spectrum of patients recruited should focus on patients who are still of working age (up to the age of 67).
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Compound score | 12 months after discharge from rehabilitation
  Compound outcome-parameter for functional recovery (from upper limb motor scores, e.g. Fugl-Meyer assessment, grip force, nine-hole peg test).

SECONDARY OUTCOMES:
Aphasia test | 3, 6 and 12 months after discharge from rehabilitation
  Standardized test for differential diagnosis Aphasia - no aphasia.
Apraxia screen of TULIA (AST) | 3, 6 and 12 months after discharge from rehabilitation
  The Apraxia Screen from TULIA is a short assessment to diagnose apraxia with 12 hand movements, dichotomous scale: 0 = not fulfilled, 1 = fulfilled motion task.
Autonomy and participation | 3, 6 and 12 months after discharge from rehabilitation
  Autonomy and participation is measured via different tools, for example with the Index for the Assessment of Health Impairments (IMET) or the subscale Participation/Role function extracted from the Stroke Impact Scale.
Fatigue scale for motor function and cognition (FSMC) | 3, 6 and 12 months after discharge from rehabilitation
  Fatigue scale for motor and cognitive functions, an assessment of fatigue, containing two subscales (mental and physical fatigue), ranging from 20 (no fatigue at all) to 100 (severest grade of fatigue).
Fugl-Meyer assessment upper extremity (FMA) | 3, 6 and 12 months after discharge from rehabilitation
  The section motor function of upper limb is one of five domains, a three-point scale is used for rating performance as 0=cannot perform, 1=performs partially and 2=performs fully, max. possible score: 66 points.
Grip and pinch force | 3, 6 and 12 months after discharge from rehabilitation
  A dynamometer is used to measure grip strength and a pinch gauge to measure pinch force.
Index for measuring restrictions on participation (IMET) | 3, 6 and 12 months after discharge from rehabilitation
  The Index of measurement of participation restrictions (IMET) records patient-related participation as a self-evaluation tool, on a scale from 0 (no impairment) to 10 (no more activity possible).
Knowledge and information needs | 3, 6 and 12 months after discharge from rehabilitation
  A questionnaire developed by the research group (including questions on informativeness and information needs on the topic of stroke).
Line bisection test (LBS) | 3, 6 and 12 months after discharge from rehabilitation
  The line bisection test (LBS) is a test to detect the presence of unilateral spatial neglect. To complete the test, the middle of several horizontal lines must be marked.
Modified Rankin Scale (MRS) | 3, 6 and 12 months after discharge from rehabilitation
  The modified Rankin scale (MRS) is a standardized measure that describes the extent of disability after a stroke. It ranges from 0 (no symptoms) to 6 (death due to stroke).
Montreal cognitive assessment (MoCA) | 3, 6 and 12 months after discharge from rehabilitation
  The Montreal Cognitive Assessment (MoCA) is a screening assessment for detecting cognitive impairment, a maximum of 30 points (no restrictions) can be achieved.
National institutes of health stroke scale (NIHSS) | 3, 6 and 12 months after discharge from rehabilitation
  The National Institutes of Health Stroke Scale, NIHSS, is a score system to quantify the impairment caused by a stroke. The sum of the values from the investigations results in a maximum of 42 points. The higher the score, the more extensive the stroke.
Nine hole peg test (NHPT) | 3, 6 and 12 months after discharge from rehabilitation
  A timed measure of fine manual dexterity where the patient is instructed to first take nine pegs out of a container and place them afterwards back into the empty holes of the container as quickly as possible.
Patient Health Questionnaire (PHQ-9) | 3, 6 and 12 months after discharge from rehabilitation
  The Patient Health Questionnaire 9 (PHQ-9) is a screening tool for diagnosing depressivity and includes questions on the nine DSM-IV criteria for the diagnosis of major depression.
Patient reported health status (EQ-5D) | 3, 6 and 12 months after discharge from rehabilitation
  The EQ-5D questionnaire is a standardized, generic measure of health-related quality of life, it is a self-administered questionnaire.
Return to work | 3, 6 and 12 months after discharge from rehabilitation
  A questionnaire developed by the research group (including questions on occupation and lifestyle).
Stroke impact scale (SIS) | 3, 6 and 12 months after discharge from rehabilitation
  Measurement of subjective stroke-specific health status, 64 items in eight domains, domain scores range between 0-100, with higher scores represent better health status.
Time up and go test (TUG) | 3, 6 and 12 months after discharge from rehabilitation
  The Timed "Up and Go" test is a clinical test to assess a patient's mobility and risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Götz Thomalla, Prof. Dr., Principal Investigator — Department of Neurology, University Medical Center Hamburg-Eppendorf; Christian Gerloff, Prof. Dr., Study Chair — Department of Neurology, University Medical Center Hamburg-Eppendorf
Locations (6):
- Germany (6):
  - Klinikum Bad Bramstedt - Klinik für Neurologische Rehabilitation, Bad Bramstedt
  - Rehaklinik Damp - Neurologie, Damp
  - Rehaklinik Geesthacht - Neurologie, Geesthacht
  - RehaCentrum Hamburg - Neurologische Rehabilitation, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Neurologie, Hamburg
  - MediClin Klinikum Soltau - Neurologische Rehabilitation, Soltau

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is planned after main publication of results.
Supporting Information: Study Protocol
Time Frame: Within 24 months after main publication.
Access Criteria: Personal login into UKE data repository.

REFERENCES:
- [Background] Birke G, Wolf S, Ingwersen T, Bartling C, Bender G, Meyer A, Nolte A, Ottes K, Pade O, Peller M, Steinmetz J, Gerloff C, Thomalla G. Protocol for a multicenter observational prospective study of functional recovery from stroke beyond inpatient rehabilitation - The Interdisciplinary Platform for Rehabilitation Research and Innovative Care of Stroke Patients (IMPROVE). Neurol Res Pract. 2020 Apr 6;2:10. doi: 10.1186/s42466-020-00056-2. eCollection 2020. PMID 33324916
- [Derived] Wolf S, Holm SE, Ingwersen T, Bartling C, Bender G, Birke G, Meyer A, Nolte A, Ottes K, Pade O, Peller M, Steinmetz J, Gerloff C, Thomalla G. Pre-stroke socioeconomic status predicts upper limb motor recovery after inpatient neurorehabilitation. Ann Med. 2022 Dec;54(1):1265-1276. doi: 10.1080/07853890.2022.2059557. PMID 35510813
- [Derived] Ingwersen T, Wolf S, Birke G, Schlemm E, Bartling C, Bender G, Meyer A, Nolte A, Ottes K, Pade O, Peller M, Steinmetz J, Gerloff C, Thomalla G. Long-term recovery of upper limb motor function and self-reported health: results from a multicenter observational study 1 year after discharge from rehabilitation. Neurol Res Pract. 2021 Dec 27;3(1):66. doi: 10.1186/s42466-021-00164-7. PMID 34955097